CLINICAL TRIAL: NCT03080649
Title: Laser in Caries Treatment - Patients´View, Pulpal Reactions and Survival of Fillings. A Randomized Controlled Trial.
Brief Title: Laser in Caries Treatment - Patients´View, Pulpal Reactions and Survival of Fillings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Dental Health in Uppsala Region (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Dr Pia Gabre, Professor, Public Dental Health in Uppsala Region
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2010/200
Record Dates: First submitted 2017-01-28; First posted 2017-03-15 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Dental Caries
Keywords: dental caries, Er:YAG laser, rotary bur
MeSH Terms: conditions — Dental Caries | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: prospective, single-blind, randomized and controlled investigation
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor have not met the patient before assessing the outcome. No information about which excavation method used is available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotary bur (Active Comparator): Device rotary bur
  Interventions: Device: excavated with rotary bur
- Er:YAG laser (Experimental): Device Er:YAG laser
  Interventions: Device: Er:YAG laser

INTERVENTIONS:
Device: excavated with rotary bur — One of two identified caries lesions in the patient were randomly allocated to be excavated with rotary bur
  Arms: Rotary bur
Device: Er:YAG laser — One of two identified caries lesions in the patient were randomly allocated to be excavated with Er:YAG laser
  Arms: Er:YAG laser

SUMMARY:
The aim of this study was to evaluate the excavation time, patients´ experiences, pulpal reactions and survival of fillings when carious tissue was removed with Er:YAG laser compared to rotary bur. A prospective, single-blind, randomized and controlled investigation was performed. Patients with at least two primary caries lesions radiographically assessed as the same size were recruited. In each patient one cavity was excavated with rotary bur and one with Er:YAG laser technique. The time requested for excavation and local anaesthesia were measured. The prevalence of postoperative symptoms, pulpal vitality and the quality of fillings will be investigated during two years after the excavation occasion.

DETAILED DESCRIPTION:
The study is a prospective, single-blind, randomized and controlled investigation. Patients between 15-40 years with at least two primary caries lesions radiographically assessed as the same size were recruited. In each patient one cavity was excavated with rotary bur and one with Er:YAG laser technique after a randomized allocation of the lesions to one of the intervention methods. The time requested for excavation to hard/firm dentin and local anaesthesia were measured. Directly after each treatment a questionnaire focusing on the experiences of the current treatment and if the laser method will be chosen in the future was answered. Postoperative pain was measured with a questionnaire one week after the treatment. Six, 12 and 24 months after the fillings were made an evaluation of pulpal status and the quality of the fillings will be performed.

ELIGIBILITY:
Inclusion Criteria:

* patients should be between 15 and 40 years,
* at least two lesions with primary caries estimated as being of equal size, and needed to be treated, in bite-wing radiographs, and
* comparable pairs of cavities should be located on either occlusal or approximal surfaces.
* the lesions should not involve the inner third of the dentin.

Exclusion Criteria:

* patients with severe general diseases ( ASA>2) (30),
* cognitive or intellectual disabilities,
* patients who required sedation or general anaesthesia, and
* teeth with periapical pathology, a root filling or non-vital teeth.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2011-08-31 (Actual); Primary Completion 2016-04-30 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Change of patients´ experience from baseline - 24 months | 0-24 months
  questionnaire

SECONDARY OUTCOMES:
Change of postoperative complications from baseline - 24 months | 0-24 months
  questionnaire
Survival of fillings | 24 months
  Registration of Ryges evaluation criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Public Dental Service, Vretgränd 9, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD are not planned to be shared